CLINICAL TRIAL: NCT05079490
Title: Impact of Motor Coordination Deficits in Preschool Children: Effects of Motor Intervention
Brief Title: Motor Intervention for Preschooler With Motor Coordination Deficits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fooyin University (Other)
Collaborators: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSVGH20-CT5-37
Record Dates: First submitted 2021-08-31; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-08

CONDITIONS: Developmental Coordination Disorder
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline (No Intervention): All children will receive outcome measures.
- Intervention phase (Experimental): Children in the experimental group will receive intervention for 12 weeks while children in the control group remain their regular activities.
  Interventions: Behavioral: motor intervention
- Follow up phase (No Intervention): All children will be followed after the end of intervention phase and receive outcome measures at 3- and 6-month after the completion of intervention.

INTERVENTIONS:
Behavioral: motor intervention — gross motor skill intervention combined with fitness training
  Arms: Intervention phase

SUMMARY:
This research project aims to examine the impact of motor coordination deficits and the effects of motor intervention on preschool-aged children's perceived competence, health-related physical fitness, activity participation and physical activity. Eighty children, aged 4-6 years,with or without motor coordination deficits will be recruited and assigned to to motor intervention (DCD-t), control 1 (DCD-c) or control 2 (TD) group. Children in the intervention group will receive motor intervention for 12 weeks. All children will be assessed at baseline, 0-, 3- and 6-month post-intervention.

DETAILED DESCRIPTION:
This research project aims to examine the impact of motor coordination deficits on preschool-aged children's perceived competence, health-related physical fitness, activity participation and physical activity. Furthermore, the investigators are to investigate the effects of motor intervention on children's competence and participation during preschool age. This study plans to recruit 40 children with motor coordination deficits, aged 4-6 years, and 40 age- and gender-matched typically developing children. Children with motor coordination deficits will further be randomly assigned to motor intervention (DCD-t) or control (DCD-c) group. At baseline assessment, all children will be assessed for motor coordination competence, self-perception of competence, health-related physical fitness and daily activity participation. Physical activity will also be quantitatively measured using accelerometry. During the intervention phase, children in the DCD-t group will receive task-oriented motor intervention combined with fitness training three times per week while children in the DCD-c group remain usual activities. All children will be re-assessed at 0-, 3- and 6-month post-intervention. Repeated Measures ANOVA will be applied to examine the differences of motor competence, self-perception, fitness and activity participation among the 3 groups of children and over the 9-month period. The effects of motor intervention on DCD children's competence and participation will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* aged 4 to 6 years
* motor coordination competence < 15%ile comparing to norms for motor-deficit group or > 30%ile for healthy group

Exclusion Criteria:

* genetic and chromosome deficits
* neurological or neuromuscular disorders
* congenital musculoskeletal disorders
* fracture in the past 6 months
* other conditions that affect the child's participation in physical activities

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
motor coordination competence- post | 3 months
  percentile scores of Movement Assessment Battery for Children, Second Edition; score range 1~99, a higher score indicates a better outcome
motor coordination competence- follow1 | 6 months
  percentile scores of Movement Assessment Battery for Children, Second Edition; score range 1~99, a higher score indicates a better outcome
motor coordination competence- follow2 | 9 months
  percentile scores of Movement Assessment Battery for Children, Second Edition; score range 1~99, a higher score indicates a better outcome
weight- post | 3 months
  body weight (kg)
weight- follow1 | 6 months
  body weight (kg)
weight- follow2 | 9 months
  body weight (kg)
height- post | 3 months
  body height (m)
height- follow1 | 6 months
  body height (m)
height- follow2 | 9 months
  body height (m)
flexibility- post | 3 months
  sit-and-reach (cm)
flexibility- follow1 | 6 months
  sit-and-reach (cm)
flexibility- follow2 | 9 months
  sit-and-reach (cm)
strength- post | 3 months
  long jump (cm)
strength- follow1 | 6 months
  long jump (cm)
strength- follow2 | 9 months
  long jump (cm)
aerobic fitness- post | 3 months
  10 meter shuttle walk test (lap)
aerobic fitness- follow1 | 6 months
  10 meter shuttle walk test (lap)
aerobic fitness- follow2 | 9 months
  10 meter shuttle walk test (lap)

SECONDARY OUTCOMES:
self-perceived motor competence- post | 3 months
  scores of Physical Competence Subscale of the The Pictorial Scale of Perceived Competence and Social Acceptance for Young Children; score range 6~24, a higher score indicates a better outcome
self-perceived motor competence- follow1 | 6 months
  scores of Physical Competence Subscale of the The Pictorial Scale of Perceived Competence and Social Acceptance for Young Children; score range 6~24, a higher score indicates a better outcome
self-perceived motor competence- follow2 | 9 months
  scores of Physical Competence Subscale of the The Pictorial Scale of Perceived Competence and Social Acceptance for Young Children; score range 6~24, a higher score indicates a better outcome
daily time spent in physical activities- post | 3 months
  7-day averaged time spent in physical activities, recorded by activity monitor (minutes per day)
daily time spent in physical activities- follow1 | 6 months
  7-day averaged time spent in physical activities, recorded by activity monitor (minutes per day)
daily time spent in physical activities- follow2 | 9 months
  7-day averaged time spent in physical activities, recorded by activity monitor (minutes per day)

CONTACTS AND LOCATIONS:
Locations (1):
- Fooyin University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No